CLINICAL TRIAL: NCT02655198
Title: Add-on Therapy With Low Dose Fenfluramine in Lennox Gastaut Epilepsy
Acronym: FFA-LGS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Collaborators: Zogenix, Inc. (Industry)
Responsible Party: Principal Investigator, Lieven Lagae, Professor Paediatric Neurology, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S58545
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Epilepsy; Lennox Gastaut Syndrome
Keywords: refractory childhood epilepsy; Lennox Gastaut syndrome; fenfluramine; anti-epileptic treatment
MeSH Terms: conditions — Epilepsy; Lennox Gastaut Syndrome | interventions — Fenfluramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fenfluramine (Experimental): Experimental : one armed open label study :
  Add-on fenfluramine in refractory Lennox Gastaut patients. Starting dose 0.2mg/kg/day. In non-responders (<50% seizure frequency decrease), dose will be uptitrated every 4 weeks from 0,2 to 0,4 and max 0,8 mg/kg/day (max 30 mg). Total duration study and max exposure to the drug 20 weeks
  Interventions: Drug: Fenfluramine

INTERVENTIONS:
Drug: Fenfluramine — study of efficacy and safety of add-on fenfluramine at different dosages in refractory Lennox Gastaut patients : 0.2 - 0.4 and 0.8 mg/kg/day (max 30 mg).

SUMMARY:
In this trial, the potential anti-epileptic effect of low dose fenfluramine in Lennox Gastaut epilepsy will be studied. An exploratory dose finding add-on trial is proposed. At baseline and at the end of the study, ECG and ultrasound of the heart will be performed as part of the safety follow up.

ELIGIBILITY:
Inclusion criteria

Electro-clinical epilepsy syndrome compatible with Lennox Gastaut syndrome:

* Minimum requirements (based on ILAE epilepsydiagnosis.org):

  * Multiple seizure types including in any case tonic seizures
  * EEG shows slow spike waves and abnormal background
  * Abnormal cognitive development
  * MRI compatible with Lennox Gastaut epilepsy : no progressive disease
* Drug resistant:

  * at least 4 documented seizures in the last 4 weeks before inclusion (minimum 4 seizures in at least 2 separate weeks) Seizure types eligible for inclusion are : generalized tonic-clonic seizures GTC , tonic seizures TS , atonic seizures AS or clearly recognizable focal seizures FS.
  * on >= 2 AEDs (including VNS) during the 4 weeks before inclusion (no changes in treatment before inclusion and during the trial)
* Age between 3 and 18 years
* Subject is male or non-pregnant, non-lactating female. Female subjects of childbearing potential must not be pregnant or breast-feeding. Female subjects of childbearing potential must have a negative urine pregnancy test. Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control, which includes abstinence, while being treated on this study and for 90 days after the last dose of study drug.

Exclusion Criteria

* Known clinical cardiovascular abnormalities (including valvular problems, shunts, pulmonary hypertension, exercise intolerance)
* Any cardiac ultrasound/ECG abnormalities at baseline
* Weight below percentile 3 for age at baseline
* Subject is receiving concomitant therapy with: centrally-acting anorectic agents; monoamine oxidase inhibitors; any centrally-acting compound with clinically appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; atomoxetine, or other centrally-acting noradrenergic agonist; cyproheptadine, and/or cytochrome P450 (CYP) 2D6/3A4/2B6 inhibitors/substrates.
* Subject is unwilling to refrain from large or daily servings of grapefruits and/or Seville oranges, and their juices beginning with the Baseline Period and throughout the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of add-on FFA in Lennox Gastaut epilepsy: Number of responders and seizure free patients at each FFA dosage (0,2 or 0,4 or 0,8 mg/kg/day) | up to 20 weeks

SECONDARY OUTCOMES:
Seizure frequency change per patient and per major seizure type (Tonic Clonic Seizures (TCS), Tonic Seizures (TS), Atonic Seizures (AS), Focal Seizures (FS)) | 20 weeks
Adverse events (cardiac and general) | 20 weeks
Sleep quality : 10 point scale instrument to score sleep quality | 20 weeks
CGI (clinical global impression) scale at last visit , by patient/caregiver and treating physician | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lieven G Lagae, MD, PhD, Principal Investigator — Katolieke Universiteit Leuven, University Hospitals Gasthuisberg
Locations (1):
- University Hospitals UZ Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Lagae L, Schoonjans AS, Gammaitoni AR, Galer BS, Ceulemans B. A pilot, open-label study of the effectiveness and tolerability of low-dose ZX008 (fenfluramine HCl) in Lennox-Gastaut syndrome. Epilepsia. 2018 Oct;59(10):1881-1888. doi: 10.1111/epi.14540. Epub 2018 Aug 26. PMID 30146701